CLINICAL TRIAL: NCT01798576
Title: Non-interventional, Observational Study on Retreatment of Chronic Hepatitis C Patients Previous Treatment Failure, Using Peginterferon Alfa-2a and Ribavirin Based Regimens
Brief Title: An Observational Study of Pegasys (Peginterferon Alfa-2a) Plus Ribavirin Based Regimens in Patients With Chronic Hepatitis C With Previous Treatment Failure
Status: Terminated | Type: Observational
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Other Study IDs: ML28498
Record Dates: First submitted 2013-02-22; First posted 2013-02-26 (Estimated); Last update posted 2016-09-15 (Estimated); Status verified 2016-09

CONDITIONS: Hepatitis C, Chronic
MeSH Terms: conditions — Hepatitis C, Chronic | interventions — peginterferon alfa-2a; Ribavirin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Pegylated interferon alfa-2a: Participants with chronic hepatitis C with previous treatment failure received combination therapy with pegylated interferon alfa-2a plus ribavirin or treatment regimens containing direct-acting anti-viral (DAAs)
  Interventions: Drug: Pegylated Interferon alfa-2a; Drug: Ribavirin

INTERVENTIONS:
Drug: Pegylated Interferon alfa-2a — Dosing was at the discretion of the investigator in accordance with local clinical practice and local labelling.
  Other Names: Peginterferon alfa 2A
Drug: Ribavirin — Dosing was at the discretion of the investigator in accordance with local clinical practice and local labelling.

SUMMARY:
This prospective, national, multicenter, observational study will evaluate in routine clinical practice the efficacy and safety of re-treatment with Pegasys (peginterferon alfa-2a) plus ribavirin or regimens containing direct-acting antivirals in participants with chronic hepatitis C who failed previous treatment. Participants will be followed for the duration of their treatment (24, 48 or 72 weeks) and for 24 weeks of follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Adult participants, >/= 18 years of age
* Participants with chronic hepatitis C who have been previously treated with pegylated interferon, standard interferon, ribavirin
* No contra-indications to pegylated interferon and ribavirin therapy or to the treatment regimen containing DAAs as detailed in the local label
* Treatment in line with summary of Product Characteristics/local labeling for Pegasys/ribavirin and DAAs, in particular:

  * Positive serum hepatitis C virus (HCV) ribonucleic acid (RNA)
  * Fertile males and females receiving ribavirin must use two forms of contraception during treatment with Pegasys/ribavirin and until 6 months post-treatment
  * No co-infection with hepatitis B or human immunodeficiency virus (HIV)

Exclusion Criteria:

* History or other evidence of a medical condition associated with chronic liver disease other than chronic hepatitis C
* History of neurological disease
* History of severe psychiatric disease
* Decompensated diabetes
* History of immunologically mediated disease
* History of severe cardiac disease
* History or evidence of severe chronic pulmonary disease
* Inadequate hematologic function
* Pregnant or breastfeeding women
* Male partners of pregnant women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Treatment-experienced participants with chronic hepatitis C receiving re-treatment with Pegasys plus ribavirin or regimens containing direct-acting antivirals (DAAs)
Sampling Method: Probability Sample
Enrollment: 282 (Actual)
Dates: Start 2012-11; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Sustained virological response (SVR) rate, defined as percentage of patients with HCV RNA <50 IU/mL at 24 weeks post completion of treatment (overall and stratified by prior treatment outcome: non-response and relapse) | approximately 3 years

SECONDARY OUTCOMES:
Percentage of patients with rapid virological response (RVR), defined as HCV RNA <50 IU/mL at Week 4 (overall and stratified by prior treatment outcome: non-response and relapse) | approximately 3 years
Percentage of patients with early virological response (EVR), defined as HCV RNA <50 IU/mL or an at least 2-log drop from baseline in HCV RNA at Week 12, but with no RVR (overall and stratified by prior treatment outcome: non-response and relapse) | approximately 3 years
Percentage of patients with non-response/relapse/virological breakthrough/virological rebound | approximately 3 years
Duration of treatment | approximately 3 years
Time to safety-related dose reduction/treatment discontinuation of any of the treatment compounds | approximately 3 years
Safety: Incidence of adverse events | approximately 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (1):
- Brasov, Romania